CLINICAL TRIAL: NCT06274879
Title: Safety of Biliary Intraductal Radiofrequency Ablation in Patients With Unresectable Extrahepatic Biliary Tract Cancer Undergoing Standard of Care Chemo-immune Checkpoint Inhibitor -Therapy: a Phase II, Multicenter, Randomized and Controlled
Brief Title: Safety of Biliary Intraductal Radiofrequency Ablation in Patients With Unresectable Extrahepatic Biliary Tract Cancer
Acronym: Ablatio
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Cancer League (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1938 Ablatio-bilica; SNCPT (Other: Portal for clinical trials in Switzerland)
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Bile Duct Cancer
Keywords: Durvalumab + chemotherapy; Radiofrequency ablation; Adverse events; Chemo-immune-checkpoint-inhibitor; Extra hepatic biliary tract cancer
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — Gemcitabine; Cisplatin; durvalumab; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Standard of care consisting of chemotherapy + durvalumab + endoscopic stenting
  Interventions: Drug: Gemcitabin, Cisplatin and Durvalumab; Procedure: Endoscopic Retrograde Cholangio-Pancreatography with stenting
- Biliary radiofrequency ablation (Experimental): Standard of care consisting of chemotherapy + durvalumab + endoscopic stenting plus intraductal radiofrequency ablation (bRFA)
  Interventions: Drug: Gemcitabin, Cisplatin and Durvalumab; Procedure: Biliary Radiofrequency Ablation; Procedure: Endoscopic Retrograde Cholangio-Pancreatography with stenting

INTERVENTIONS:
Drug: Gemcitabin, Cisplatin and Durvalumab — CICI (Gemcitabin d1 & d8 Cisplatin d1 & d8, Durvalumab d1) are administered repeating every 21 days for a total of 8 cycles.
Procedure: Biliary Radiofrequency Ablation — Biliary Radiofrequency Ablation is applied at baseline, 6 and 12 weeks
  Arms: Biliary radiofrequency ablation
Procedure: Endoscopic Retrograde Cholangio-Pancreatography with stenting — ERCP with stenting are applied at baseline and as clinically indicated

SUMMARY:
The goal of this clinical trial is to provide evidence for the general tolerability of radiofrequency ablation (bRFA) in patients with unresectable bile duct cancer undergoing systemic palliative treatment consisting of chemotherapy (gemcitabine and cisplatin) plus durvalumab (immune-checkpoint-inhibitor, ICI). The main question it aims to answer is whether it is safe to combine chemotherapy (gemcitabine and cisplatin) and immunotherapy (durvalumab) - CICI therapy.

Participants will be assigned to either the control group or the experimental group. In the control group, the standard of care consists of endoscopy with stent placement in the bile duct and CICI, whereas in the experimental group, bRFA will be performed in addition to the standard of care. Participants will be followed up for 6 months, during the follow-up, the stage of the tumor, blood examination, the duration of the stent from the insertion until its failure, adverse events and quality of life will be examined.

Researchers will compare the standard of care alone to the experimental group to see if the additional bRFA procedure causes higher or no difference in adverse events rate.

DETAILED DESCRIPTION:
Extrahepatic biliary tract cancer (EBTC) in most cases is diagnosed at an unresectable stage of disease. Standard-of-care systemic palliative treatment consists of chemotherapy (gemcitabine and cisplatin) plus durvalumab (immune-checkpoint-inhibitor, ICI). Nonetheless, overall survival remains limited at about 12.8 months. Moreover, severe adverse events can occur leading to treatment discontinuation increasing the risk of tumor progression and poor prognosis. Biliary obstruction is one of the most relevant factors for survival limiting eligibility and timing/dosing of chemo-immunotherapy. Endoscopic biliary stenting is standard to relieve jaundice, but tumor ingrowth can limit the rate and duration of success. Radiofrequency ablation (RFA) results from thermal damage created by a high-frequency alternating current released from an electrode into tissue. RFA has become a standard treatment modality in numerous indications, including the treatment of Barrett's oesophagus-related dysplasia and hepatocellular carcinoma. Intraductal biliary radiofrequency ablation (bRFA) is a relatively new method of inducing tumor necrosis via thermal energy. bRFA has been applied in patients suffering unresectable EBTC within randomized-controlled trials indicating improved stent patency as well as overall survival and progression-free survival.

The primary objective of the study is to provide evidence for the general tolerability of bRFA in patients with unresectable extrahepatic biliary tract cholangiocarcinoma undergoing CICI. It is hypothesis that bRFA is generally safe and well tolerated by patients. Primary endpoint of the study is any grade 3 or 4 adverse events leading to chemo-immune checkpoint inhibitor-therapy discontinuation up to six months after enrolment.

Eligible patients will be registered in the study database and randomized in 1:2 ratio to either the standard group (CICI with endoscopic biliary stenting) or the experimental bRFA group (CICI with endoscopic biliary stenting + bRFA).

CICI with endoscopic biliary stenting are standard of care applied commonly in both the control and the experimental group:

Endoscopic retrograde cholangiography (ERC) procedure stenting are applied at baseline and as clinically indicated. CICI cycle (Gemcitabin d1 & d8, Cisplatin d1 & d8, Durvalumab d1) are administered repeating every 21 days for a total of 8 cycles.

bRFA will be applied only to the experimental group, it is standardized as for generator settings and protocol adapting to tumor morphology using the probe at baseline, 6 and 12 weeks after study start.

ELIGIBILITY:
Inclusion criteria

1. Male or female ≥18 years old.
2. Histologically or cytologically confirmed diagnosis of previously untreated and unresectable*, locally advanced and/or metastatic extrahepatic biliary tract cholangiocarcinoma with obstructive jaundice (increased serum level of total bilirubin).
3. ECOG performance status 0 to 1.
4. Adequate bone marrow function: Neutrophil count ≥1.0 x 109/L, platelet count ≥100 x 109/L.
5. Adequate renal function: Estimated Glomerular Filtration Rate (eGFR) ≥50mL/min/1.73m2.
6. Willing and able to provide written informed consent. *The reason for inoperability needs to be documented and categorized as follows: - Locally advanced or vascular invasion = surgically not removable. - Distant metastasis.

   * Severe comorbidities.
   * Other reasons. Exclusion criteria

<!-- -->

1. Solely intrahepatic cholangiocarcinoma or mixed type liver tumors (cholangiocarcinoma with hepatocellular differentiation parts).
2. Multiple hepatic metastases with significant blockage of one or more liver segments and/or less than 50% of liver parenchyma potentially drainable on pre-intervention imaging.
3. Received prior systemic treatment for unresectable and/or metastatic Extrahepatic Biliary Tract Cancer (EBTC).
4. Any autoimmune diseases including inflammatory disorders such as Crohn's disease, ulcerative colitis, Wegener granulomatosis, systemic lupus erythematosus, rheumatoid arthritis, Graves' disease.

   Exceptions:
   * Hypothyroidism following Hashimoto thyroiditis stable on hormone replacement.
   * Patients with vitiligo.
   * Any chronic skin disorders that do not require systemic treatment.
5. Use of immunosuppressive medication within 3 weeks prior to the dose of durvalumab.

   Exceptions:

   - Topical or inhaled steroids.

   - Systemic corticosteroids at physiologic doses not exceeding >10mg/d of prednisone or equivalent.
6. Known history of Human Immunodeficiency Virus.
7. Prior Self-Expandable Metal Stent (SEMS) placement.
8. Biliary obstruction of non-tumoral etiology.
9. Liver cirrhosis Child-Pugh B or C.
10. Platelets <100 x 109/L or International Normalised Ratio (INR) >1.5.
11. History of organ transplantation.
12. Secondary tumor.

Exceptions:

- Tumor treated with curative intent without recurrence for more than 5 years.

* Non-melanoma skin cancer treated carcinoma in situ without evidence of disease. 14. Other concomitant disease or condition likely to significantly decrease life expectancy i.e., life expectancy is less than 3 months according to investigator judgement.

  15. Pregnancy or lactation. A negative blood or urine pregnancy test must be available before administration of CICI.

  16. Known or suspected non-compliance, drug, or alcohol abuse. 17. Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the candidate.

  18. Participation in another interventional study within 30 days prior to enrollment.

  19. Previous participation in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Any grade 3 or 4 adverse events (AE) leading to chemo-immune checkpoint inhibitor-therapy (CICI) discontinuation up to six months after randomization. | 6 months
  AEs will be assessed according to US National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v5). Treatment discontinuation is defined as deferral of administration by at least four weeks or a definite stop of all CICI agents.

SECONDARY OUTCOMES:
Endoscopic complications as measured by the Adverse events GastRointestEstinal Endoscopy (AGREE) criteria specifically developed for endoscopic interventions | 6 months
  Current guideline definitions for cholangitis, post-ERCP pancreatitis and bleeding are applied. The rate of readmissions for biliary complications will be assessed specifically by being defined as any non-elective endoscopic reintervention after the first stent placement and will be documented in terms of timing, type of intervention, hospitalization and its duration and resolution.
Progression-free survival: The time until either progression of the underlying disease or death, whichever occurs first, assessed from the time of up to 6 months after randomization. | 6 months
Death from any cause at the follow-up at 6 months after randomization (overall survival). | 6 months
Disease-specific quality-of-life as measured by the EORTC QLQ-BIL21 before every CICI cycle and at 3 and 6 months after the start of CICI treatment. | 6 months
  EORTC QLQ-BIL21 (European Organisation for Research and Treatment of Cancer questionnaire for measuring quality of life in patients with cholangiocarcinoma and cancer of the gallbladder), scores range from 0 to 100, where a lower score means a better quality of life.
Change in health-related quality-of-life at baseline, 3 and 6 months from the start of the CICI treatment as measured by the EORTC QLQ-C30 | 6 months
  EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer questionnaire quality of life questionnaire core 30), scores range from 0 to 100, where a high scale score represents a higher response level.
Stent patency at month 3 visit and at 6 months after the start of CICI treatment. | 6 months
Number of courses of CICI applied | 6 months
Total dose of CICI applied | 6 months
Number of patients with any grade 3 or 4 Adverse Events (AE) leading to discontinuation or non-initiation of CICI up to six months after randomization. | 6 months
Number of patients not starting CICI within 4 weeks after randomization. | 6 months
Time from randomization to CICI start. | 6 months

OTHER OUTCOMES:
Details of adverse events | 6 months
Overall survival at 24 months after randomization | 24 months
  This will be an investigator-initiated sub-study outside this protocol

CONTACTS AND LOCATIONS:
Overall Officials: Reiner Prof. Dr. med. Wiest, Principal Investigator — Inselspital Bern University Hospital
Locations (1):
- Inselspital Bern University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
This will be planned only at study completion

REFERENCES:
- [Background] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Background] Rimini M, Fornaro L, Lonardi S, Niger M, Lavacchi D, Pressiani T, Lucchetti J, Giordano G, Pretta A, Tamburini E, Pirrone C, Rapposelli IG, Diana A, Martinelli E, Garajova I, Simionato F, Schirripa M, Formica V, Vivaldi C, Caliman E, Rizzato MD, Zanuso V, Nichetti F, Angotti L, Landriscina M, Scartozzi M, Ramundo M, Pastorino A, Daniele B, Cornara N, Persano M, Gusmaroli E, Cerantola R, Salani F, Ratti F, Aldrighetti L, Cascinu S, Rimassa L, Antonuzzo L, Casadei-Gardini A. Durvalumab plus gemcitabine and cisplatin in advanced biliary tract cancer: An early exploratory analysis of real-world data. Liver Int. 2023 Aug;43(8):1803-1812. doi: 10.1111/liv.15641. PMID 37452505